CLINICAL TRIAL: NCT01090518
Title: Cortisol Augmentation of a Psychological Treatment in Warfighters With Post Traumatic Stress Disorder (PTSD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Collaborators: Lightfighter Trust (Unknown)
Responsible Party: Principal Investigator, Rachel Yehuda, PhD, Professor of Neuroscience and Psychiatry, Bronx VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LFT2009-02-1
Record Dates: First submitted 2010-03-11; First posted 2010-03-22 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged Exposure therapy with Hydrocortisone (Active Comparator)
  Interventions: Behavioral: Prolonged Exposure therapy; Drug: Hydrocortisone
- Prolonged Exposure therapy with placebo (Placebo Comparator)
  Interventions: Behavioral: Prolonged Exposure therapy

INTERVENTIONS:
Behavioral: Prolonged Exposure therapy — 10 weekly sessions
  Arms: Prolonged Exposure therapy with Hydrocortisone
Drug: Hydrocortisone — 30mg 20 minutes prior to each PE session including imaginal exposure (8 total)
  Arms: Prolonged Exposure therapy with Hydrocortisone
Behavioral: Prolonged Exposure therapy — 10 weekly sessions
  Arms: Prolonged Exposure therapy with placebo

SUMMARY:
This study seeks to examine the efficacy of hydrocortisone administration in the augmentation of the therapeutic effects of Prolonged Exposure (PE) therapy, an empirically tested treatment shown to be effective in the the treatment of posttraumatic stress disorder (PTSD). The augmentation builds on both the translation of neuroscience findings demonstrating the effects of glucocorticoids (GCs) on learning, and on empirical clinical findings from other investigators demonstrating beneficial effects of GCs in reducing traumatic memories in trauma-exposed persons.

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of chronic PTSD according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnostic criteria, resulting from a deployment-related traumatic event, and a minimum PTSD severity of 50 (CAPS).
* The veteran must either be unmedicated or on a stable psychotropic regimen (i.e., 1 or more months on the same regimen).

Exclusion Criteria:

* Lifetime history of psychotic disorder, bipolar disorder, or obsessive compulsive disorder.
* Moderate or severe traumatic brain injury (TBI).
* A medical or mental health problem other than PTSD that requires immediate clinical attention.
* Substance abuse or dependence within the last 3 months.
* Suicidal risk (as determined by response of 5 or 6 on the suicidality items of the Montgomery Asberg Depression Rating Scale (MADRS)) and/or assessed suicide risk on the basis of clinical judgment.
* Persons on a psychotropic medication regimen that has not been consistent for one month.
* Presence of diabetes mellitus or any current unstable medical illness or condition that represents a contraindication to taking glucocorticoids (this will be determined by history and/or abnormal laboratory findings at medical clearance).
* Unwillingness to discontinue other specialized psychotherapy for PTSD during the 10 weeks of study treatment and the 6 week follow-up. (Self-help (non-trauma focused) groups or supportive counseling can be continued but not initiated.)
* Pregnant women or those planning to become pregnant within the study period will not be enrolled. Female participants must agree to use an effective method of birth control (i.e., oral contraceptive, Norplant, diaphragm, condom, or spermicide, abstinence) during the course of the study to ensure they do not become pregnant during the course of the study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
PTSD symptom severity as assessed by the Clinician Administered PTSD Scale (CAPS) | week 0
PTSD symptom severity as assessed by the Clinician Administered PTSD Scale (CAPS) | week 10
PTSD symptom severity as assessed by the Clinician Administered PTSD Scale (CAPS) | week 16

SECONDARY OUTCOMES:
Cognitive performance (learning and retention in an episodic memory task, attention and working memory) | week 0
Cognitive performance (learning and retention in an episodic memory task, attention and working memory) | week 10
Cognitive performance (learning and retention in an episodic memory task, attention and working memory) | week 16
Other measures of clinical outcome, psychological state and functioning | week 0
Other measures of clinical outcome, psychological state and functioning | week 10
Other measures of clinical outcome, psychological state and functioning | week 16
Biological measures associated with PTSD severity | week 0
Biological measures associated with PTSD severity | week 10
Biological measures associated with PTSD severity | week 16

CONTACTS AND LOCATIONS:
Locations (1):
- James J. Peters Veterans Affairs Medical Center, The Bronx, New York, United States